CLINICAL TRIAL: NCT00003809
Title: Randomized, Double Blind, Placebo Controlled Phase III Evaluation of Cisplatin + Placebo Versus Cisplatin + C225 a Mouse/Human Monoclonal Antibody to the Epidermal Growth Factor Receptor, in Patients With Metastatic and/or Recurrent Squamous Cell Cancer of the Head and Neck
Brief Title: Cisplatin With or Without Monoclonal Antibody Therapy in Treating Patients With Metastatic or Recurrent Head and Neck Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066954; ECOG-E5397
Record Dates: First submitted 1999-11-01; First posted 2004-04-14 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Head and Neck Cancer
Keywords: untreated metastatic squamous neck cancer with occult primary; recurrent metastatic squamous neck cancer with occult primary; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab; Cisplatin

INTERVENTIONS:
Biological: cetuximab
Drug: cisplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies can locate cancer cells and either kill them or deliver tumor-killing substances to them without harming normal cells. It is not yet known whether cisplatin plus monoclonal antibody therapy is more effective than cisplatin alone for metastatic or recurrent head and neck cancer.

PURPOSE: Randomized double-blinded phase III trial to compare the effectiveness of cisplatin with or without monoclonal antibody in treating patients who have metastatic or recurrent head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the efficacy (survival and response rates) and toxicity of cisplatin with or without monoclonal antibody C225 in patients with metastatic and/or recurrent squamous cell head and neck cancer. II. Compare the correlation between epidermal growth factor receptor density and response and progression-free survival in these patients. III. Determine the steady state serum levels of monoclonal antibody C225 and the frequency of human antibody response to this monoclonal antibody in patients treated with the combination therapy.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients are stratified according to disease status (newly diagnosed vs recurrent) and ECOG status (0 vs 1). Patients are randomized to 1 of 2 treatment arms. Arm I: Patients receive monoclonal antibody C225 IV over 2 hours followed 1 hour later by cisplatin IV over 2 hours on day 1 of course 1. Monoclonal antibody C225 is administered over 1 hour on subsequent courses. Arm II: Patients receive placebo IV over 2 hours followed 1 hour later by cisplatin as in arm I on day 1 of course 1. Placebo is administered over 1 hour on subsequent courses. Treatment continues every 4 weeks for at least 6 courses in the absence of disease progression or unacceptable toxicity. Arm II patients who develop disease progression may then crossover to arm I treatment. Patients are followed at 1 and 3 months and then every 3 months until disease progression.

PROJECTED ACCRUAL: A total of 114 patients will be accrued for this study within 14 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven squamous cell carcinoma of the head and neck that is incurable with surgery or radiotherapy No nasopharyngeal primaries Measurable or evaluable disease Newly diagnosed with extensive, incurable local regional disease AND distant metastases OR Local regional recurrence/persistence or distant metastases after surgery or radiotherapy Persistent or progressive disease after radiotherapy must be histologically proven at least 8 weeks after therapy No brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 10 g/dL (transfusion allowed) Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT and SGPT no greater than 2 times upper limit of normal (ULN) Alkaline phosphatase no greater than 2 times ULN Renal: Creatinine no greater than 1.2 mg/dL OR Creatinine clearance at least 50 mL/min Calcium no greater than ULN No history of hypercalcemia Other: No active infection No other concurrent malignancy within past 2 years except curatively treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix No known hypersensitivity to murine proteins Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior chimeric antibody or kinase inhibitor for recurrent or metastatic disease No more than 1 prior biotherapy regimen for recurrent or metastatic disease Chemotherapy: At least 3 months since prior induction or adjuvant chemotherapy concurrent with radiotherapy No prior chemotherapy for recurrent disease Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics At least 4 weeks since prior radiotherapy Surgery: See Disease Characteristics Recovered from prior major surgery

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-08-06 (Actual); Primary Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara A. Burtness, MD, Study Chair — Yale University
Locations (76):
- United States (73):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Beckman Research Institute, City of Hope, Los Angeles, California
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - Stanford University Medical Center, Stanford, California
  - CCOP - Colorado Cancer Research Program, Inc., Denver, Colorado
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Gainsville, Gainesville, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Veterans Affairs Medical Center - Tampa (Haley), Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - New England Medical Center Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Riverview Medical Center, Red Bank, New Jersey
  - St. Francis Medical Center, Trenton, New Jersey
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Veterans Affairs Medical Center - New York, New York, New York
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Ireland Cancer Center, Cleveland, Ohio
  - Veterans Affairs Medical Center - Cleveland, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Sooner State, Tulsa, Oklahoma
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Penn State Geisinger Cancer Center, Hershey, Pennsylvania
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Veterans Affairs Medical Center - Pittsburgh, Pittsburgh, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - Veterans Affairs Medical Center - Nashville, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Medical Research and Education Foundation, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
- Puerto Rico (2):
  - MBCCOP - San Juan, San Juan
  - Veterans Affairs Medical Center - San Juan, San Juan
- Pretoria Academic Hospitals, Pretoria, South Africa

REFERENCES:
- [Result] Burtness B, Goldwasser MA, Flood W, Mattar B, Forastiere AA; Eastern Cooperative Oncology Group. Phase III randomized trial of cisplatin plus placebo compared with cisplatin plus cetuximab in metastatic/recurrent head and neck cancer: an Eastern Cooperative Oncology Group study. J Clin Oncol. 2005 Dec 1;23(34):8646-54. doi: 10.1200/JCO.2005.02.4646. PMID 16314626
- [Result] Burtness BA, Li Yi, Flood W, et al.: Phase III trial comparing cisplatin (C) + placebo (P) to C + anti-epidermal growth factor antibody (EGF-R) C225 in patients (pts) with metastatic/recurrent head & neck cancer (HNC). [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-901, 2002.
- [Derived] Chung CH, Lee JW, Slebos RJ, Howard JD, Perez J, Kang H, Fertig EJ, Considine M, Gilbert J, Murphy BA, Nallur S, Paranjape T, Jordan RC, Garcia J, Burtness B, Forastiere AA, Weidhaas JB. A 3'-UTR KRAS-variant is associated with cisplatin resistance in patients with recurrent and/or metastatic head and neck squamous cell carcinoma. Ann Oncol. 2014 Nov;25(11):2230-2236. doi: 10.1093/annonc/mdu367. Epub 2014 Jul 31. PMID 25081901